CLINICAL TRIAL: NCT05303272
Title: A Crossover, Randomized and Multi-center Study to Evaluate the Efficacy and Safety of Abatacept Versus Mycophenolate Mofetil (MMF) in Treatment of PV
Brief Title: A Study to Evaluate Efficacy and Safety of Abatacept in Participants of Pemphigus Vulgaris (PV)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Wuhan Central Hospital (Other); Wuhan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, YIKAI YU, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TJRH2021109
Record Dates: First submitted 2022-02-25; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus | interventions — Abatacept; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abatacept (Experimental): Subject received subcutaneous administration of abatacept 125 mg once every week through the 52 week double blind period.
  Interventions: Drug: Abatacept Prefilled Syringe
- Mycophenolate mofetil (Active Comparator): Subject received subcutaneous administration of matching placebo of abatacept once a weeks through the 24 week double blind period. A washout period of MMF for 4 weeks (24 th-28th week) is used to ensure data integrity. Subsequently,subject were administered subcutaneous administration of abatacept 125 mg once every week through the 28-52 week open label period.
  Interventions: Drug: Mycophenolate Mofetil 500Mg Tab

INTERVENTIONS:
Drug: Abatacept Prefilled Syringe — Abatacept (Orencia) was provided in prefilled glass syringes initial syringes contained 0.6ml (60mg) of concentration 100 mg/m: drug product subsequently modified to 0.4 mL (20mg) concentration (50mg/ML) drug product. Combined with standard of care prednisone 10-40mg qd
  Other Names: Orencia
  Arms: Abatacept
Drug: Mycophenolate Mofetil 500Mg Tab — MMF will be administered at a starting dose of 1000 milligrams (mg) Q12H and the dose will be tapered to achieve a goal of 0.5-1.0 gram (gm) Q12H. Combined with standard of care prednisone 10-40mg qd through 52 weeks.
  Other Names: MMF,CellCept
  Arms: Mycophenolate mofetil

SUMMARY:
Pemphigus vulgaris (PV) is a rare, chronic, debilitating, and potentially life-threatening autoimmune disorder that is characterized by mucocutaneous blisters.Abatacept is a biologic drug that belongs to the class of T-cell co-stimulation modulators and is used for the treatment of autoimmune diseases.

DETAILED DESCRIPTION:
The background therapy is based on prednisolone administration. PV is a rare disorder, therefore this study is designed as a crossover that may require fewer patients than a parallel study. The study enrolled participants with moderate-to-severely active PV requiring ≥ 50 milligrams per day (mg/day) oral prednisone or equivalent. The purpose of this study was to evaluate the efficacy, tolerability, and safety of abatacept injection for subcutaneous use (abatacept SC) 150 mg administered once in a week in subjects with PV. It was anticipated that with sustained immune suppression in the presence of abatacept SC that clinical remission of the disease would be improved.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 through 80 years of age) with clinically-documented diagnosis of PV for >2 months and <10 years.
2. History of biopsy consistent with PV (Hematoxylin and Eosin staining and direct immunofluorescence). Confirmed diagnosis of PV within the previous 24 months, based on the presence of histological features of acantholysis via skin or mucosal biopsy and one of the following: tissue bound immunoglobulin G (IgG) antibodies by direct immunofluorescence on the surface of affected epithelium or serological detection of serum desmoglein-3 (DSg3) autoantibodies against epithelial cell surface either by indirect immunofluorescence microscopy or by enzyme-linked immunosorbent assay.
3. At least 1 previous episode of a failed steroid taper (ie, disease flare/relapse) at a prednisone/prednisolone dose >10 mg/day. The following criteria must have been met as evidence of disease severity at the time of the failed steroid taper: a) A Pemphigus Severity of Clinical Disease score of moderate (2) or severe (3) (may be historical/retrospective assessment). b) Required a treatment change at the time of the failed steroid taper of at least one of the following: i) A steroid increase to >=20 mg/day OR ii) The addition of immunosuppressive/immunomodulatory agent/treatment OR iii) A dose increase of immunosuppressive/immunomodulatory agent/treatment
4. Screening anti-Dsg antibodies consistent with a diagnosis of PV (ie, elevated antiDsg3 antibodies).
5. Has initiated and received a stable dose of prednisone/prednisolone from a minimum of 20 mg/day (example: 0.25 mg/kg/day for an 80 kg person) up to a maximum of 120 mg/day or 1.5 mg/kg/day (whichever is higher) for >=2 weeks prior to randomization.
6. Has exhibited PV disease control, defined as no new lesions for >=2 weeks. A female subject is eligible to enter the study if she: Is of non-child bearing potential, who 7. is either surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or post-hysterectomy) or is postmenopausal without menses for >2 years. Women who are <2 years postmenopausal are required to have menopausal status confirmed by follicle-stimulating hormone (FSH) and estradiol levels at the screening evaluation. If FSH and estradiol levels do not provide confirmation of menopause, subject will be considered to be of childbearing potential.

Exclusion Criteria:

1. Diagnosis of pemphigus foliaceus, paraneoplastic pemphigus, or other autoimmune blistering disease (other than pemphigus vulgaris).
2. Past or current history of hypersensitivity to components of the investigational product or medically significant adverse effects (including allergic reactions) from cetirizine (or antihistamine equivalent) or paracetamol/acetaminophen.
3. Prior treatment with rituximab without achieving disease control within 6 months of initiating rituximab dosing.
4. Prior treatment with immunosuppressant or immunomodulation agents within the protocol specified periods
5. Evidence or history of clinically significant infections
6. Past or current malignancy, except for cervical carcinoma Stage 1B or less, noninvasive basal cell and squamous cell skin carcinoma and cancer diagnoses with a duration of complete response (remission) >5 years
7. Significant concurrent, uncontrolled medical condition that could affect the subject's safety, impair the subject's reliable participation in the study, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol. This includes subjects who require any systemic steroid treatment for a concurrent medical condition (other than pemphigus vulgaris).
8. Use of an investigational drug or other experimental therapy within 4 weeks, 5 pharmacokinetic half-lives, or the duration of biological effect (whichever is longer) prior to Screening.
9. Electrocardiogram (ECG) showing a clinically significant abnormality or showing a QTc interval ≥450 msec (≥480 msec for subjects with a bundle branch block)
10. Woman who is breastfeeding.
11. Positive test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV) serology at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Achieved Sustained Complete Remission, Evaluated by the Pemphigus Disease Area Index (PDAI) Activity Score | 24 Weeks
  PADAI and ABSIS was proposed by the German Blistering Disease Group in 2007 which was accepted as the most sensitive and reliable systems for evaluation of pemphigus severity. PADAI was developed by the International Pemphigus Definitions Group in 2009
Percentage of Participants Who Achieved Sustained Complete Remission, Evaluated byAutoimmune bullous skin disorder intensity score (ABSIS) | 24 Weeks
  PADAI and ABSIS was proposed by the German Blistering Disease Group in 2007 which was accepted as the most sensitive and reliable systems for evaluation of pemphigus severity. PADAI was developed by the International Pemphigus Definitions Group in 2009

SECONDARY OUTCOMES:
Cumulative Oral Corticosteroid Dose | From 12th, 24th, 36th and 52th Week
  Calculate the Cumulative Oral Corticosteroid Dose during 52 week
Ulcer Severity Score (USS) for the assessment of skin, oral ulcer improvement | From baseline up to 4th, 8th,12th, 24th, 36th and 52th Week
  The USS incorporates six ulcer characteristics: number, size, duration, ulcer-free period, site, and pain. This scoring template may be of value to future studies assessing treatment efficacy.
Physician global assessment (PGA) | From baseline up to 4th, 8th,12th, 24th, 36th and 52th Week
  Physician global assessment was assessed by an individual researcher
Autoimmune bullous disease quality of life (ABQoL) | From baseline up to 4th, 8th,12th, 24th, 36th and 52th Week
  Total ABQoL scores range from 0 to 30 with higher DLQI scores reflecting greater impairment in a participant's health-related quality of life. The ABQoL score is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The measure type mean is the estimated mean from adjusted MMRM.
Anti-desmoglein 1 (anti-Dsg1) and anti-Dsg3 autoantibody titers | From Baseline up to 12th, 24th and 52th Week
  anti-Dsg1 and anti-Dsg3 will be performed using ELISA
Change From Baseline for CD19+ B Cell Count | From Baseline up to 12th, 24th and 52th Week
  CD19+ B cell count will be performed using Flow Cytometry

CONTACTS AND LOCATIONS:
Overall Officials: AIHUA DU, M.D, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No